CLINICAL TRIAL: NCT02452138
Title: Endotoxin Activity Assay and Microcirculation Examination in Patients With Severe Sepsis
Brief Title: Endotoxin Activity Assay and Microcirculation in Severe Sepsis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201503015RINB
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Low EAA: Endotoxin Activity Assay [EAA] level < 0.40 EAA units
  Interventions: Other: Severe sepsis management
- Intermediate EAA: Endotoxin Activity Assay [EAA] level between 0.40-0.59 EAA units
  Interventions: Other: Severe sepsis management
- High EAA: Endotoxin Activity Assay [EAA] level >= 0.60 EAA units
  Interventions: Other: Severe sepsis management

INTERVENTIONS:
Other: Severe sepsis management

SUMMARY:
Endotoxin is the major mediator of sepsis resulted from systemic inflammatory response syndrome induced by gram-negative bacteria infection. The endotoxin related inflammatory response and hypercoagulation can result in microcirculatory dysfunction. When microcirculatory dysfunction is severe, it can induce multiple organ dysfunction syndrome and death. This is a prospective observational study, and it will not influence the sepsis treatment decision of the medical care team. The critically ill severe sepsis patients will be enrolled only if they meet all inclusion criteria, do not meet any exclusion criteria and sign the consent form after explanation of the aim and process of the trial by the primary investigator or research personnel. After enrollment, the patient will receive serum assay of endotoxin activity (EAA) and endocan level. The patient will also receive examination of sublingual microcirculation by using the incident dark field video microscope. After 24 hours, the patient will receive assay of endocan level and examination of sublingual microcirculation. This study will record the vital signs, laboratory data, dose of vasopressors and inotropic agents, and severity of organ dysfunction. After 28 days, this study will check the survival, stay of intensive care, stay of hospital, ventilator day, and the results of culture of pathogens. The patients will be assign to the following three groups by the EAA level: low EAA group (< 0.40 EAA units); intermediate EAA group (0.40-0.59 EAA units); and high EAA group (≧ 0.60 EAA units). This grouping will be used for statistical analysis and comparison. The primary goal of this study is to investigate the difference of the prevalence of gram-negative bacteria infection, pathogen, infection source, microcirculation, the severity of disease, and the prognosis among these three groups.

ELIGIBILITY:
Inclusion Criteria:

* patients with the following infections: intraabdominal infection, pneumonia, urinary tract infection, blood stream infection, or wound infection
* patients must also meet any one of the following criteria for severe sepsis

  * SBP < 90 mm Hg, MAP < 65 mm Hg, or requirement of vasopressors or inotropics
  * PaO2/FiO2 < 300
  * Creatinine level > 2 mg/dL or increase > 0.5 mg/dL; or urine output < 0.5 mL/kg/h more than 2 hours
  * Bilirubin level > 4 mg/dL
  * Platelet count < 100 k/uL or decrease more than 50%
  * INR > 1.5 or aPTT > 60 sec
  * GCS < 13 or 9T
  * Lactate > 2 mmol/L (with pH < 7.3 or base excess < -5 mmol/L)

Exclusion Criteria:

* younger than 20 yeras old or greater than 99 years old
* the onset of severe sepsis before enrollment is greater than 24 hours
* pregnant
* have received plymyxin-B hemoperfusion within 24 hours before enrollment
* non-native speaker

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe sepsis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-05 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Difference of the prevalence of gram-negative bacteria infection | At enrollment
  Compare the prevalnce of gram-negative bacteria infection among the three groups

SECONDARY OUTCOMES:
Difference of Total small vessel density | At Enrollment
  Total small vessel density will be measured by incident dark field video microscope. Compare the difference among the three groups.
Difference of Perfused small vessel density | At enrollment
  Perfused small vessel density will be measured by incident dark field video microscope. Compare the difference among the three groups.
Endocan level | At enrollment
  Endocan level will be measured by Human Endocan kit. Compare the difference among the three groups.
SOFA score | At enrollement
  Compare the Sequential Organ Failure Assessment score among the three groups
28-day mortality | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chang Yeh, MD, PhD, Principal Investigator — National Taiwan University Hospital